CLINICAL TRIAL: NCT06022042
Title: Clinical Comparison of On1 Two-stage Abutment With One-stage Abutment on Different Implant Neck Design
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Zhou (Other)
Responsible Party: Sponsor-Investigator, Yi Zhou, Deputy Chief Physician, Deputy Director of Dental Implant Department, The Dental Hospital of Zhejiang University School of Medicine
Organization: The Dental Hospital of Zhejiang University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHZhejiangU-2022(027)
Record Dates: First submitted 2022-03-09; First posted 2023-09-01 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Implant Site Reaction

STUDY DESIGN:
Intervention Model Description: The researchers prospectively and continuously recruited subjects who underwent implant therapy in the Oral Implantation Center of the Stomatology Hospital Affiliated to Zhejiang University School of Medicine, and all subjects who signed written informed consent were divided into 8 groups by random number table method: ① On1 abutment + Nobel Replace Conical Connection PMC implant group (hereinafter referred to as Nobel PMC), ②On1 abutment + Nobel Parallel™ Conical Connection implant group (hereinafter referred to as Nobel PCC), ③On1 abutment + Nobel Replace Conical Connection implant group (Hereinafter referred to as Nobel CC), ④ One-stage abutment + Nobel PMC implant set, ⑤ One-stage abutment + Nobel PCC implant set, ⑥ One-stage abutment + Nobel CC implant set.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study takes a single-blind method. During research process, the researchers cannot avoid knowing the type of abutment used by the subjects during the clinical examination and operation, so the subjects can only be single-blinded.The clinical examination data were measured and averaged by two independent clinicians. The data was analysed by a third person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- On1 Abutment + Nobel PMC implant Set (Experimental): Subjects who takes implant therapy using On1 Abutment + Nobel PMC implant
  Interventions: Device: On1 two-stage abutment and one-stage abutment
- On1 Abutment + Nobel PCC Implant Set (Experimental): Subjects who takes implant therapy using On1 Abutment + Nobel PCC Implant
  Interventions: Device: On1 two-stage abutment and one-stage abutment
- On1 Abutment + Nobel CC Implant Set (Experimental): Subjects who takes implant therapy using On1 Abutment + Nobel CC Implant
  Interventions: Device: On1 two-stage abutment and one-stage abutment
- One-Stage Abutment + Nobel PMC Implant Set (Active Comparator): Subjects who takes implant therapy using One-Stage Abutment + Nobel PMC Implant
  Interventions: Device: On1 two-stage abutment and one-stage abutment
- One-Stage Abutment + Nobel PCC Implant Set (Active Comparator): Subjects who takes implant therapy using One-Stage Abutment + Nobel PCC Implant
  Interventions: Device: On1 two-stage abutment and one-stage abutment
- One-Stage Abutment + Nobel CC Implant Set (Active Comparator): Subjects who takes implant therapy using One-Stage Abutment + Nobel CC Implant
  Interventions: Device: On1 two-stage abutment and one-stage abutment

INTERVENTIONS:
Device: On1 two-stage abutment and one-stage abutment — the On1 two-stage abutment has a smooth collar with a height of 1.75-2.5mm, and the Nobel implants have a smooth neck design ranging from 0-0.75mm to protect the connective tissue around the implant.
  Other Names: Nobel PMC implant, Nobel CC implant, Nobel PCC implant

SUMMARY:
In clinical implant treatment, the healing abutment or temporary abutment needs to be removed or replaced multiple times after implant insertion and before prosthesis restoration. During this process, the friction between connective tissue around the implant cannot be avoided. Different from natural periodontal tissue, soft tissue around the implant lacks the periodontal ligament barrier and periodontal ligament blood supply, and is more likely to be damaged during repeated wearing. The integrity, health and stability of the peri-implant connective tissue is crucial to the implant osseointegratio. Through randomized controlled trials and meta-analysis, Marco Tallarico et al found that repeated removal of one-stage abutments can significantly increase bone resorption.

Based on this situation, the design of implant neck and abutment, especially the design concept of smooth collar, has attracted widespread attention. The design of smooth collars with different heights can isolate the mechanical damage of the abutment to the connective tissue around the implant to different degrees. Among them, the On1 two-stage abutment has a smooth collar with a height of 1.75-2.5mm, and the Nobel implants have a smooth neck design ranging from 0-0.75mm to protect the connective tissue around the implant. Through a systematic review and meta-analysis, Qing-qing Wang et al concludes that direct mechanical stimulation from the abutment has long-term adverse effects on peri-implant connective tissue and bone tissue. However, whether the On1 two-stage abutment has a positive effect on the stabilization of the peri-implant soft tissue and bone tissue remains to be studied.

At the same time, the relative height of the smooth collar increased by the On1 abutment in the implants with different neck designs varies to some extent, and further research is still needed to provide evidence about the effect of the On1 abutment on the tissue surrounding the implants with different neck designs. In conclusion, this study took On1 two-stage abutment and traditional one-stage abutment as the research objects to compare and evaluate the clinical effects of the two in different implant neck design.

DETAILED DESCRIPTION:
Research purpose To compare the clinical effects of On1 two-stage abutment and one-stage abutment in implants with different neck design.

Research Design and Methods

1. Type of study design: prospective intervention single-center randomized clinical trial
2. Study period: 7 years
3. Start time: from the date of ethics approval, end time: March 2029
4. This study takes a single-blind method. During research process, the researchers cannot avoid knowing the type of abutment used by the subjects during the clinical examination and operation, so the subjects can only be single-blinded.

Measures to control bias:

1. Selection bias control: use the random number table method for grouping, and strictly follow the blinding method. During the recruiting period, the researcher needs to fully know the subjects and improve the understanding and compliance of the test; during the recruiting period, at least 2 contact information should be left. In emergencies, the subjects themselves can be contacted to minimize the rate of loss to follow-up; for those fail to follow-up, data will be excluded in the follow-up statistical phase;
2. Control of information bias: 1) rigorously design case report forms, 2) set up two 3) Collect data on objective indicators as much as possible, conduct regular researcher training, and unify evaluation standards;
3. Control confounding bias: improve the study design, control single variable grouping, and adopt reasonable statistical analysis methods.

5. Subject inclusion criteria, exclusion criteria, and withdrawal criteria

Inclusion criteria:

(1) aged 18 years and above, 70 years old and below; (2) Single crown restoration after implantation (3) Subjects signed written informed consent; (4) The general health status is good and adhered to Good oral hygiene conditions; (5) no infection and extraction residues at the implant site; (6) sufficient keratinized gingiva on the cheek and tongue; (7) good and stable occlusal relationship; (8) the occlusal gap is higher than 4mm; (9) No other additional operations are planned to perform.

Exclusion criteria:

(1) contraindications to general implant surgery; (2) uncontrolled diabetes mellitus; (3) any signs of immunosuppression; (4) previous head and neck radiation therapy; (5) past or current use of bisphosphonates treatment; (6) substance abuse; (7) nocturnal teeth grinding; (8) signs of periodontitis; (9) smoking more than 10 cigarettes per day; (10) poor oral hygiene; (11) mental disorders; (12) inability to complete follow-up; (13) History of night grinding.

Withdrawal criteria:

(1) abnormal vital organ function (2) poor compliance (3) serious adverse reactions (4) poor efficacy (5) intolerance of adverse reactions (6) willing to take other treatment methods or withdraw without any reason.

6. Design plan and expected duration and specific arrangements for participating in clinical trials: Subjects are expected to participate in clinical trials for 7 years, and need to complete follow-up. Imaging examinations, including parallel projection X-rays and CBCT, are required on the day of surgery, 3 months, 6 months, and 1-7 years after surgery.

7. Trial suspension criteria: According to the clinical trial protocol, ① Controllable adverse events occur, or safety problems are found, which can be reasonably controlled by improving the research design or means. Suspend and adjust clinical trial protocols in a timely manner. ② Some subjects could not avoid the influence of specific risks, so the trial was suspended in time and susceptible subjects were excluded. ③ The data obtained are extremely statistically significant. Apply for an interim analysis.

Criteria for termination of the trial: ① There are serious adverse events, and the adverse events are likely to be related to the intervention in the trial; ② External information (such as other high-quality research or evidence) proves that the intervention is ineffective or effective, and the current clinical trial is not necessary to continue, ③ According to the planned interim analysis to achieve the expected difference in efficacy, if it has been observed that the intervention program of the experimental group is significantly better than that of the control group.

Statistical analysis: The homogeneity of variance is planned to be tested within groups, the outcome indicators of different groups are planned to be analyzed by variance between groups, and further correlation analysis is planned to perform on indicators with significant differences.

8. The clinical observations, clinical examination values, imaging measurements, and clinical scale scores generated by the investigator's examination in this study, and original records were made. The source data record shall indicate the record time, record source and recorder.

9. Main outcome measures: buccal bone wall thickness at 0/2/4/6 mm below the implant shoulder; The degree of bone resorption at the shoulder edge of the implant, the distance between the level of implant shoulder and the alveolar ridge.

Secondary observation indicators: mesial and distal gingival papilla and buccal mucosa recession; abutment buccal keratinized gingiva width; probing bleeding index; Red aesthetic index, subject self-satisfaction, and time to subsidence of mucous membrane blushing when wearing teeth.

10. The specific research plan is as follows: The researchers prospectively and continuously recruited subjects who underwent implant therapy in the Oral Implantation Center of the Stomatology Hospital Affiliated to Zhejiang University School of Medicine, and all subjects who signed written informed consent were divided into 8 groups by random number table method: ① On1 abutment + Nobel Replace Conical Connection PMC implant group (hereinafter referred to as Nobel PMC), ②On1 abutment + Nobel Parallel™ Conical Connection implant group (hereinafter referred to as Nobel PCC), ③On1 abutment + Nobel Replace Conical Connection implant group (Hereinafter referred to as Nobel CC), ④ One-stage abutment + Nobel PMC implant set, ⑤ One-stage abutment + Nobel PCC implant set, ⑥ One-stage abutment + Nobel CC implant set. The subjects' basic information, clinical and imaging findings were collected. Complete preoperative examinations and records were carried out before surgery. Immediately postoperatively, the width of the buccal keratinized gingiva of the healing abutment was recorded and examined by imaging. Clinical examinations were performed 1 week, 3 months, 4 months, 6 months, and 1-7 years after surgery, including: mesial and distal gingival papilla and buccal mucosa recession, and the width of the buccal keratinized gingiva of the abutment. Among them, regular imaging examinations, including parallel projection X-rays and CBCT, were performed immediately after surgery, 3 months after surgery, and 1-7 years after surgery. Only small dental radiographs were taken 6 months after the operation.

Sample Size Calculation

The sample size of this study was estimated by G*Power software. To satisfy statistical significance, set the conditions as t tests, α=0.05, 1-β=0.9. Referring to studies of the same type [3], the effect size ES f=0.8 was set, and the minimum sample size of each group was calculated to be 28. Based on the standard of 5% loss to follow-up rate, the number of subjects recruited in each group of this study is set to be 30. The grouping design and sample size are as follows:

group design sample size On1 abutment + Nobel PMC implant set, 30 On1 Abutment + Nobel PCC Implant Set 30 On1 Abutment + Nobel CC Implant Set 30 One-Stage Abutment + Nobel PMC Implant Set 30 One-Stage Abutment + Nobel PCC Implant Set 30 One-Stage Abutment + Nobel CC Implant Set 30 Data management and confidentiality

1. The clinical examination data were measured and averaged by two independent clinicians, recorded in the case collection form, and analyzed by a third person using spss19.0 statistical software to evaluate whether there were statistical differences. The imaging data were called and analyzed by submitting an application to the Affiliated Stomatology Hospital of Zhejiang University School of Medicine. During the process, the patient's real name was hidden, and the data quality assurance management was carried out according to the following requirements: ① Exclude all missing data, unused data and illogical data. 2) Screening and sorting out the test data that meet the inclusion criteria, forming a data set of observational safety and various clinical effects and conducting statistical analysis.
2. Modification procedure for deviation from the original statistical analysis plan: submit a deviation report form to the ethics committee. In addition to the deviation statement, the table shows the frequency of each type of deviation and its impact on the research results. Behavior is explained and there are actions taken for deviations from the plan.
3. All records related to the identity of the subjects are kept confidential, and these materials will not be disclosed to the public outside the scope permitted by relevant laws and/or regulations.

Informed consent This study will be conducted by the research doctor in the Oral Implantation Center of Zhejiang University Affiliated Stomatology Hospital, and the subjects will be informed and informed consent will be obtained before surgery. The informed consent process conforms to the principles of complete notification, full understanding, and independent choice; the expression of informed consent is easy to understand and conforms to the level of understanding of the subject group.

This study does not involve vulnerable groups. All subjects will sign the informed consent form by themselves.

Adverse event reporting This study did not include measures and interventions other than routine clinical treatment, and had no other adverse effects on the subjects.

In the event of an adverse event, we will report it as follows:

Various adverse events: Take timely measures to deal with them and record them in the case report form.

Serious adverse events (SAE): take measures to deal with them timely, and record in a case report form, stop the trial at the decision of the investigator, immediately report to the ethics committee, drug clinical trial institutions and sponsors, and report to national and provincial food within 24 hours Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 18 years and above, 70 years old and below; (2) Single crown restoration after implantation (3) Subjects signed written informed consent; (4) The general health status is good and adhered to Good oral hygiene conditions; (5) no infection and extraction residues at the implant site; (6) sufficient keratinized gingiva on the cheek and tongue; (7) good and stable occlusal relationship; (8) the occlusal gap is higher than 4mm; (9) No other additional operations are planned to perform.

Exclusion Criteria:

* (1) contraindications to general implant surgery; (2) uncontrolled diabetes mellitus; (3) any signs of immunosuppression; (4) previous head and neck radiation therapy; (5) past or current use of bisphosphonates treatment; (6) substance abuse; (7) nocturnal teeth grinding; (8) signs of periodontitis; (9) smoking more than 10 cigarettes per day; (10) poor oral hygiene; (11) mental disorders; (12) inability to complete follow-up; (13) History of night grinding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
The degree of bone resorption at the shoulder edge of the implant | 1-7 years
  1. Thickness of the buccal bone plate 0 mm below the implant abutment (W1): Select the mid-axis of the implant in the sagittal plane.The thickness of the lateral buccal plate (W1) is determined by selecting the mid-axis of the implant in the sagittal plane and making a straight line perpendicular to the long axis of the implant to the buccal side of the implant table.
  2. Thickness of the buccal bone plate 2、4、6 mm below the implant abutment (W2、W3、W4): select the sagittal implant centre axis and make a straight line perpendicular to the long axis of the implant, starting from the buccal bone plate.(W2、W3、W4): Choose the mid-axis of the implant in the sagittal plane and start from the buccal bone plate and make a straight line perpendicular to the long axis of the implant to the distance from the buccal side of the implant 2、4、6 mm below the shoulder table.
The distance between the level of implant shoulder and the alveolar ridge. | 1-7 years
  The distance between the level of implant shoulder and the alveolar ridge.

SECONDARY OUTCOMES:
buccal bone wall thickness at 0/2/4/6 mm below the implant shoulder | 1-7 years
  1. Level of the implant at the top of the proximal mesial alveolar ridge (HM): selecting the coronal implant mesial axis, the distance from the proximal mesial alveolar crest to the horizontal line of the implant abutment.
  2. Level of the implant at the top of the distal mesial alveolar ridge (HD): Selection of the coronal implant mesial axis, distance from the top of the distal mesial alveolar ridge to the implant abutment level.The distance from the top of the crest to the horizontal line of the implant abutment.
  3. Level of the implant at the apex of the buccal alveolar ridge (HB): distance from the apex of the buccal alveolar ridge to the level of the implant abutment, with the implant in the sagittal plane selected for the medial axis.
mesial and distal gingival papilla and buccal mucosa recession | 1-7 years
  mesial and distal gingival papilla and buccal mucosa recession
abutment buccal keratinized gingiva width | 1-7 years
  abutment buccal keratinized gingiva width
probing bleeding index | 1-7 years
  probing bleeding index
Patients' self-satisfaction visual analogue scale score | within 30 minutes
  Patients were also assessed by visual anlog scale (VAS) for The degree of pain and self-satisfaction of wearing the teeth was assessed using the visual anlog scale (VAS) [11]. A 10 cm long scale with the leftmost end scored as 0 means no pain (unsatisfactory); the rightmost end scored as 0 means no pain (unsatisfactory); the rightmost end scored as 0 means no pain (unsatisfactory); and the rightmost end scored as 0 means no pain (unsatisfactory). (unsatisfactory); the right-most end of the scale was scored as 10, indicating severe pain (extremely satisfactory). The patient marks the scale according to his/her own feelings. The patient marks the scale according to his/her own feelings, with 1cm representing 1 point, and the indicated position is converted into the final score.
time to subsidence of mucous membrane blushing when wearing teeth | within 30 minutes
  time to subsidence of mucous membrane blushing when wearing teeth

CONTACTS AND LOCATIONS:
Overall Officials: Weida Li, Principal Investigator — Stomatological Hospital Affiliated to Zhejiang University School of Medicine
Locations (1):
- The Stomatologic Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tallarico M, Caneva M, Meloni SM, Xhanari E, Covani U, Canullo L. Definitive Abutments Placed at Implant Insertion and Never Removed: Is It an Effective Approach? A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Oral Maxillofac Surg. 2018 Feb;76(2):316-324. doi: 10.1016/j.joms.2017.08.025. Epub 2017 Aug 24. PMID 28923270
- [Background] Wang QQ, Dai R, Cao CY, Fang H, Han M, Li QL. One-time versus repeated abutment connection for platform-switched implant: A systematic review and meta-analysis. PLoS One. 2017 Oct 19;12(10):e0186385. doi: 10.1371/journal.pone.0186385. eCollection 2017. PMID 29049323